CLINICAL TRIAL: NCT01798394
Title: Progesterone & Postpartum Relapse to Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012NTLS059; R21DA034840 (NIH)
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder
Keywords: pregnant; smoker; cigarette; tobacco
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Active Comparator): Take micronized natural progesterone capsule by mouth, twice daily (approximately at 8 am and 8 pm) for four weeks beginning on postpartum day 4.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): Take placebo capsule by mouth, twice daily (approximately at 8 am and 8 pm) for 4 weeks beginning on postpartum day 4.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Progesterone — Take micronized natural progesterone capsule by mouth, twice daily (approximately at 8 am and 8 pm) for four weeks beginning on postpartum day 4.
  Other Names: Prometrium
  Arms: Progesterone
Other: Placebo — Take placebo capsule by mouth, twice daily (approximately at 8 am and 8 pm) for 4 weeks beginning on postpartum day 4.
  Arms: Placebo

SUMMARY:
The primary goal of this project is to investigate the potential efficacy of exogenous progesterone (with supplemental relapse prevention counseling) on postpartum relapse in new mothers. Also to determine the feasibility of enhanced compliance monitoring and identification of collateral factors effecting outcomes.

DETAILED DESCRIPTION:
Pregnant women will be recruited at gestational weeks 33-36 who have quit smoking during pregnancy and are motivated to maintain abstinence after delivery. At the time of delivery, women will be randomly assigned to receive 4 weeks of active or placebo exogenous progesterone starting on the 4th day postpartum. Participants will be in contact with study staff either by phone or clinic visits until 12 weeks postpartum to collect data on smoking status and protocol compliance, measure serum progesterone levels and receive behavioral counseling.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* 18-35 years old
* Zero CPD for past 4 weeks
* 5 or more CPD for at least 6 out of past 12 months
* Motivated to remain abstinent (7 or higher out of 10)
* Stable physical/mental health
* Established prenatal care
* Stable physical/mental health
* Willing to take Progesterone
* Willing to use double-barrier protection if sexually active
* English fluency
* Able to provide informed consent

Exclusion Criteria:

* Psychotropic medications
* Illicit drugs
* Other types of tobacco, NRT, smoking cessation medications
* Pregnancy complications (Diabetes, Anomaly, Fetal growth restriction, HTN, Hx of >2 miscarriages)
* Current use of: Finasteroid (propecia), Efavirenz, Red Clover, Ketoconazole, CYP3A4 Inhibitors
* History of: Thrombophelitis, Deep vein thrombosis, Pulmonary embolus, Clotting disorder, Bleeding disorder, Heart disease, Diabetes, Stroke, Peanut allergy, Liver dysfunction, Hypersensitivity to progesterone

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon S. Allen, M.D., Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota, 717 Delaware Street SE, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Progesterone | Placebo
Started | 24 | 22
Completed | 21 | 19
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone | Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.5) | 26.7 (5.0) | 26.5 (5.2)
Gender [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Relapsed by Week 4 Postpartum
Description: Determined by seven-day point prevalence, a binary smoking relapse outcome - defined as a single puff of a cigarette during the seven days prior to a pre-specified time point of interest.
Time Frame: Week 4 Postpartum
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 24 | 22
participants | 6 | 7

2. Secondary Outcome: Number of Participants Who Relapsed by Week 12 Postpartum
Description: as for outcome 1
Time Frame: Week 12 Postpartum
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 24 | 22
participants | 11 | 13

3. Secondary Outcome: Number of Participants Who Relapsed at All During Postpartum (up to Day 84)
Description: Defined by continuous abstinence (CA) defined as a single puff of a cigarette as a relapse.
Time Frame: Postpartum Day 0 to 84
Measure: Number; unit: participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 24 | 22
participants | 10 | 13

4. Secondary Outcome: Protocol Compliance - Number of Visits Attended
Description: Compliance was measured as the number of visits attended (maximum of 5).
Time Frame: Gestational Week 36 - Postpartum Week 12
Measure: Mean (Standard Deviation); unit: Number of visits attended
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 24 | 22
Number of visits attended | 4.5 (1.1) | 4.4 (1.2)

5. Secondary Outcome: Compliance Determinants
Description: This was determined by the Feasibility Questionnaire; a 10-item measure used to assess participant expectations, satisfaction of study protocol, study medication and electronic data capture. All questions were answered on a four-point Likert-type scale (1=low acceptability and 4=high acceptability). The total score was determined by adding up all the scores and dividing by 10.
Time Frame: Postpartum Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 24 | 22
units on a scale | 3.6 (0.3) | 3.5 (0.3)

6. Secondary Outcome: Protocol Compliance - Doses of Medication Taken
Description: Compliance was measured by doses of medication taken (maximum of 56).
Time Frame: Postpartum Week 0 - Week 12
Measure: Mean (Standard Deviation); unit: Doses of medication taken
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 24 | 22
Doses of medication taken | 38.9 (22.3) | 37.5 (18.3)

7. Secondary Outcome: Protocol Compliance - EDC's Completed
Description: Compliance was measured as the number by number of EDCs completed (maximum of 84).
Time Frame: Gestational Week 36 - Postpartum Week 12
Measure: Mean (Standard Deviation); unit: EDC's completed
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 24 | 22
EDC's completed | 60.9 (21.8) | 61.8 (24.3)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Progesterone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=24) | Placebo (N=22)
Hospitalization for post-cesarean section infection (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes